CLINICAL TRIAL: NCT03578965
Title: Does Antibiotic Prophylaxis Reduce Wound Complications After Vulvar Excision of Premalignant Lesions: A Double-Blinded Randomized Controlled Trial
Brief Title: Does Antibiotic Prophylaxis Reduce Wound Complications After Vulvar Excision of Premalignant Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201804136
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Results first posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Premalignant Vulvar Lesion; Benign Vulvar Lesion
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The principal investigator along with all members of the study team involved in data analysis as well as the patients will be blinded to the randomization group. The research assistant will disclose the randomization group to the anesthesiologist who will screen the patient for allergies and then obtain the appropriate antibiotics from the pharmacy and administer the antibiotics as appropriate. These will be administered prior to the procedure and so the surgeon will remain blinded to the administration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: No antibiotic prophylaxis prior to skin incision (No Intervention): -Women randomized to no antibiotic prophylaxis will not receive any antibiotics prior to skin incision.
- Arm B: Antibiotic prophylaxis prior to skin incision (Experimental): -Women randomized to prophylactic antibiotics will receive a cefazolin as per ACOG guidelines.
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — -If patient has a penicillin allergy then clindamycin will be used. Prophylactic antibiotics should be administered prior to skin incision
  Arms: Arm B: Antibiotic prophylaxis prior to skin incision

SUMMARY:
A randomized control trial will provide the most reliable data to determine the role of prophylactic antibiotics to decrease the wound complication rate. The investigators plan to perform a pilot study to evaluate actual rates of wound complications and how long it takes to recruit 50 patients.

ELIGIBILITY:
Inclusion Criteria:

* All women, >=18 undergoing vulvar surgery
* Biopsy proven benign or premalignant lesion requiring surgical management.
* Women of childbearing age will be required to have a negative human chorionic gonadotropin (HCG) test within seven days of surgery.
* Scheduled to undergo surgical management for their vulvar disease supervised by a faculty member within the Division of OBGYN at Washington University School of Medicine
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Women who are pregnant
* Women scheduled to undergo a radical vulvectomy
* Women scheduled to undergo a concomitant graft, flap or plastic surgery
* Women <18 years of age
* History of prior vulvar radiation
* Inability to sign an informed consent form prior to registration on study
* Inability to understand spoken or written English
* Prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Mullen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (10.3) | 56.1 (14.4) | 53.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 26 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 9 | 11
  White | 21 | 17 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50
Diagnosis of diabetes mellitus [Count of Participants; unit: Participants] | 1 | 8 | 9
Diagnosis of HIV [Count of Participants; unit: Participants] | 0 | 1 | 1
Immunosuppressive medications [Count of Participants; unit: Participants] | 1 | 0 | 1
Steroid use [Count of Participants; unit: Participants] | 2 | 0 | 2
Diagnosis of hypertension [Count of Participants; unit: Participants] | 6 | 18 | 24
Diagnosis of congestive heart failure [Count of Participants; unit: Participants] | 0 | 1 | 1
Diagnosis of cardiac valvular disease [Count of Participants; unit: Participants] | 0 | 6 | 6
Diagnosis of coronary artery disease [Count of Participants; unit: Participants] | 1 | 4 | 5
Diagnosis of chronic kidney disease [Count of Participants; unit: Participants] | 3 | 6 | 9
Diagnosis of pulmonary disease [Count of Participants; unit: Participants] | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Vulvar Wound Complications Compared Between the Two Arms
Description: Wound complication will be defined as a composite outcome that includes wound breakdown, sterile site infection, hematoma, seroma diagnosed within 30 days after excision. Sterile Site Infection (SSI) - defined as purulent drainage, cellulitis, abscess, or a wound that requires drainage, debridement or antibiotics associated with a clinical diagnosis of infection.
Time Frame: Within 30 days of surgery (estimated to be 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
Number analyzed (Participants) | 24 | 26
Participants | 6 | 10

2. Secondary Outcome: Clinical Risk Factors That Correlate With Vulvar Wound Complications as Measured by Demographic Variables That Predispose Patients to Infection
Description: Clinical risk factors could include history of diabetes, liver disease, human immunodeficiency virus, chronic kidney disease, congestive heart failure, chronic obstructive pulmonary disease, peripheral vasculature disease, dementia, connective tissues disease, leukemia, lymphoma, peptic ulcer disease, hypertension, steroid use, and use of other immunosuppressive medications.
Time Frame: Within 30 days of surgery (estimated to be 30 days)
Population: The number analyzed for each row equals the number of participants who had the listed pre-existing condition or medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
Number analyzed (Participants) | 24 | 26
Participants
  HIV: number analyzed (Participants) | 0 | 1
  HIV: Vulvar wound complication(s) | 0 | 0
  HIV: No vulvar wound complication(s) | 0 | 1
  Immunosuppressive medications: number analyzed (Participants) | 1 | 0
  Immunosuppressive medications: Vulvar wound complication(s) | 0 | 0
  Immunosuppressive medications: No vulvar wound complication(s) | 1 | 0
  Steroid use: number analyzed (Participants) | 2 | 0
  Steroid use: Vulvar wound complication(s) | 0 | 0
  Steroid use: No vulvar wound complication(s) | 2 | 0
  Diabetes mellitus: number analyzed (Participants) | 1 | 8
  Diabetes mellitus: Vulvar wound complication(s) | 0 | 2
  Diabetes mellitus: No vulvar wound complication(s) | 1 | 6
  Hypertension: number analyzed (Participants) | 6 | 18
  Hypertension: Vulvar wound complication(s) | 1 | 5
  Hypertension: No vulvar wound complication(s) | 5 | 13
  Congestive heart failure: number analyzed (Participants) | 0 | 1
  Congestive heart failure: Vulvar wound complication(s) | 0 | 0
  Congestive heart failure: No vulvar wound complication(s) | 0 | 1
  Cardiac valvular disease: number analyzed (Participants) | 0 | 6
  Cardiac valvular disease: Vulvar wound complication(s) | 0 | 3
  Cardiac valvular disease: No vulvar wound complication(s) | 0 | 3
  Coronary artery disease: number analyzed (Participants) | 1 | 4
  Coronary artery disease: Vulvar wound complication(s) | 0 | 1
  Coronary artery disease: No vulvar wound complication(s) | 1 | 3
  Chronic kidney disease: number analyzed (Participants) | 3 | 6
  Chronic kidney disease: Vulvar wound complication(s) | 0 | 2
  Chronic kidney disease: No vulvar wound complication(s) | 3 | 4
  Pulmonary disease: number analyzed (Participants) | 5 | 12
  Pulmonary disease: Vulvar wound complication(s) | 2 | 4
  Pulmonary disease: No vulvar wound complication(s) | 3 | 8

3. Secondary Outcome: Association of Postoperative Vulvar Hygiene Adherence With Vulvar Wound Complications
Description: * Patients will complete the Vulvar Hygiene Survey 2-3 weeks post surgery.
  * The after surgery section asks 6 questions about if the patient performed specific vulvar hygienic procedures
Time Frame: Within 30 days of surgery (estimated to be 30 days)
Population: The number analyzed in the rows below do not match the overall number of participants analyzed in some categories because the participant did not answer the question on the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
Number analyzed (Participants) | 24 | 26
Participants
  Chose to not sit and to lie/stand when possible = yes: number analyzed (Participants) | 21 | 16
  Chose to not sit and to lie/stand when possible = yes: Vulvar wound complication(s) | 5 | 8
  Chose to not sit and to lie/stand when possible = yes: No vulvar wound complication(s) | 16 | 8
  Chose to not sit and to lie/stand when possible = no: number analyzed (Participants) | 3 | 8
  Chose to not sit and to lie/stand when possible = no: Vulvar wound complication(s) | 1 | 2
  Chose to not sit and to lie/stand when possible = no: No vulvar wound complication(s) | 2 | 6
  Regularly performed vulvar wound care = yes postop: number analyzed (Participants) | 22 | 23
  Regularly performed vulvar wound care = yes postop: Vulvar wound complication(s) | 5 | 10
  Regularly performed vulvar wound care = yes postop: No vulvar wound complication(s) | 17 | 13
  Regularly performed vulvar wound care = no: number analyzed (Participants) | 1 | 1
  Regularly performed vulvar wound care = no: Vulvar wound complication(s) | 0 | 0
  Regularly performed vulvar wound care = no: No vulvar wound complication(s) | 1 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times a day postop for 1-2 days: number analyzed (Participants) | 3 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times a day postop for 1-2 days: Vulvar wound complication(s) | 0 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times a day postop for 1-2 days: No vulvar wound complication(s) | 3 | 0
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 3-7 days: number analyzed (Participants) | 0 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 3-7 days: Vulvar wound complication(s) | 0 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 3-7 days: No vulvar wound complication(s) | 0 | 0
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 8-14 days: number analyzed (Participants) | 9 | 3
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 8-14 days: Vulvar wound complication(s) | 5 | 2
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 8-14 days: No vulvar wound complication(s) | 4 | 1
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 14+ days: number analyzed (Participants) | 6 | 11
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 14+ days: Vulvar wound complication(s) | 1 | 4
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for 14+ days: No vulvar wound complication(s) | 5 | 7
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for unknown # of days: number analyzed (Participants) | 2 | 0
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for unknown # of days: Vulvar wound complication(s) | 0 | 0
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop for unknown # of days: No vulvar wound complication(s) | 2 | 0
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop = no: number analyzed (Participants) | 4 | 8
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop = no: Vulvar wound complication(s) | 0 | 2
  Performed sitz baths or cleansed with a showerhead 2-3 times per day postop = no: No vulvar wound complication(s) | 4 | 6
  Actively kept the vulva dry postop 1-2 days: number analyzed (Participants) | 0 | 0
  Actively kept the vulva dry postop 1-2 days: Vulvar wound complication(s) | 0 | 0
  Actively kept the vulva dry postop 1-2 days: No vulvar wound complication(s) | 0 | 0
  Actively kept the vulva dry postop 3-7 days: number analyzed (Participants) | 2 | 4
  Actively kept the vulva dry postop 3-7 days: Vulvar wound complication(s) | 0 | 2
  Actively kept the vulva dry postop 3-7 days: No vulvar wound complication(s) | 2 | 2
  Actively kept the vulva dry postop 8-14 days: number analyzed (Participants) | 11 | 7
  Actively kept the vulva dry postop 8-14 days: Vulvar wound complication(s) | 4 | 2
  Actively kept the vulva dry postop 8-14 days: No vulvar wound complication(s) | 7 | 5
  Actively kept the vulva dry postop 14+ days: number analyzed (Participants) | 6 | 11
  Actively kept the vulva dry postop 14+ days: Vulvar wound complication(s) | 1 | 4
  Actively kept the vulva dry postop 14+ days: No vulvar wound complication(s) | 5 | 7
  Actively kept the vulva dry postop for unknown # of days: number analyzed (Participants) | 2 | 0
  Actively kept the vulva dry postop for unknown # of days: Vulvar wound complication(s) | 0 | 0
  Actively kept the vulva dry postop for unknown # of days: No vulvar wound complication(s) | 2 | 0
  Actively kept the vulva dry postop = no: number analyzed (Participants) | 3 | 2
  Actively kept the vulva dry postop = no: Vulvar wound complication(s) | 1 | 0
  Actively kept the vulva dry postop = no: No vulvar wound complication(s) | 2 | 2
  Cleaned the vulva after urinating postop 1-2 days: number analyzed (Participants) | 0 | 0
  Cleaned the vulva after urinating postop 1-2 days: Vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after urinating postop 1-2 days: No vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after urinating postop 3-7 days: number analyzed (Participants) | 2 | 4
  Cleaned the vulva after urinating postop 3-7 days: Vulvar wound complication(s) | 0 | 4
  Cleaned the vulva after urinating postop 3-7 days: No vulvar wound complication(s) | 2 | 0
  Cleaned the vulva after urinating postop 8-14 days: number analyzed (Participants) | 10 | 6
  Cleaned the vulva after urinating postop 8-14 days: Vulvar wound complication(s) | 3 | 1
  Cleaned the vulva after urinating postop 8-14 days: No vulvar wound complication(s) | 7 | 5
  Cleaned the vulva after urinating postop 14+ days: number analyzed (Participants) | 10 | 12
  Cleaned the vulva after urinating postop 14+ days: Vulvar wound complication(s) | 3 | 4
  Cleaned the vulva after urinating postop 14+ days: No vulvar wound complication(s) | 7 | 8
  Cleaned the vulva after urinating postop for unknown # of days: number analyzed (Participants) | 1 | 1
  Cleaned the vulva after urinating postop for unknown # of days: Vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after urinating postop for unknown # of days: No vulvar wound complication(s) | 1 | 1
  Cleaned the vulva after urinating postop = no: number analyzed (Participants) | 1 | 2
  Cleaned the vulva after urinating postop = no: Vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after urinating postop = no: No vulvar wound complication(s) | 1 | 2
  Cleaned the vulva after having a bowel movement postop 1-2 days: number analyzed (Participants) | 0 | 0
  Cleaned the vulva after having a bowel movement postop 1-2 days: Vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after having a bowel movement postop 1-2 days: No vulvar wound complication(s) | 0 | 0
  Cleaned the vulva after having a bowel movement postop 3-7 days: number analyzed (Participants) | 3 | 4
  Cleaned the vulva after having a bowel movement postop 3-7 days: Vulvar wound complication(s) | 0 | 3
  Cleaned the vulva after having a bowel movement postop 3-7 days: No vulvar wound complication(s) | 3 | 1
  Cleaned the vulva after having a bowel movement postop 8-14 days: number analyzed (Participants) | 10 | 5
  Cleaned the vulva after having a bowel movement postop 8-14 days: Vulvar wound complication(s) | 3 | 1
  Cleaned the vulva after having a bowel movement postop 8-14 days: No vulvar wound complication(s) | 7 | 4
  Cleaned the vulva after having a bowel movement postop 14+ days: number analyzed (Participants) | 9 | 10
  Cleaned the vulva after having a bowel movement postop 14+ days: Vulvar wound complication(s) | 3 | 4
  Cleaned the vulva after having a bowel movement postop 14+ days: No vulvar wound complication(s) | 6 | 6
  Cleaned the vulva after having a bowel movement postop for unknown # of days: number analyzed (Participants) | 1 | 1
  Cleaned the vulva after having a bowel movement postop for unknown # of days: Vulvar wound complication(s) | 0 | 1
  Cleaned the vulva after having a bowel movement postop for unknown # of days: No vulvar wound complication(s) | 1 | 0
  Cleaned the vulva after having a bowel movement postop = no: number analyzed (Participants) | 1 | 3
  Cleaned the vulva after having a bowel movement postop = no: Vulvar wound complication(s) | 0 | 1
  Cleaned the vulva after having a bowel movement postop = no: No vulvar wound complication(s) | 1 | 2

4. Secondary Outcome: Incidence of Adverse Events to Antibiotic Use
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: Within 30 days of surgery (estimated to be 30 days)
Population: Only participants in Arm B who received antibiotic prophylaxis are evaluable for this outcome measure
Measure: Number; unit: adverse events
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
Number analyzed (Participants) | 0 | 26
adverse events |  | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days after completion of study treatment (estimated to be 31 days)
Arm/Group | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision | Arm B: Antibiotic Prophylaxis Prior to Skin Incision
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 20/24 | 17/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: No Antibiotic Prophylaxis Prior to Skin Incision (N=24) | Arm B: Antibiotic Prophylaxis Prior to Skin Incision (N=26)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hemorrhoid (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Minimal pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Swollen sensation (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vulvar infection (Infections and infestations) | 0 | 1
Bloody discharge (Injury, poisoning and procedural complications) | 0 | 1
Discolored suture (Injury, poisoning and procedural complications) | 0 | 1
Easy bruising (Injury, poisoning and procedural complications) | 1 | 0
Vulvar bleeding (Injury, poisoning and procedural complications) | 1 | 0
Vulvar discomfort (Injury, poisoning and procedural complications) | 1 | 0
Vulvar wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Vulvar wound drainage (Injury, poisoning and procedural complications) | 1 | 2
Vulvar/vaginal discharge (Injury, poisoning and procedural complications) | 4 | 1
Vulvar/vaginal spotting (Injury, poisoning and procedural complications) | 1 | 1
Wound separation (Injury, poisoning and procedural complications) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Mood changes (Psychiatric disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Pain with intercourse (Reproductive system and breast disorders) | 0 | 1
Vaginal bleeding (Reproductive system and breast disorders) | 1 | 0
Vulvar pain (Reproductive system and breast disorders) | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Arm and thigh itching (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1
Vulvar pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Vulvar rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03578965/Prot_SAP_000.pdf